CLINICAL TRIAL: NCT06987565
Title: Transcutaneous Vagus Nerve Stimulation in SLE (TvSSLE)
Brief Title: Transcutaneous Vagus Nerve Stimulation in SLE
Acronym: TvSSLE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Lupus Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-0331
Record Dates: First submitted 2025-04-23; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Pain; Vagus nerve stimulation
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus Nerve Stimulation (Active Comparator): Patients will receive transcutaneous stimulation of the left vagus nerve for 5 minutes daily for 28 consecutive days.
  Interventions: Device: Active vagus nerve stimulation
- Sham Vagus Nerve Stimulation (Placebo Comparator): Patients will receive sham transcutaneous stimulation of the of the left vagus nerve for 5 minutes daily for 28 consecutive days.
  Interventions: Device: Sham vagus nerve stimulation

INTERVENTIONS:
Device: Active vagus nerve stimulation — Patients will receive transcutaneous stimulation of the vagus nerve for 5 minutes daily for 28 consecutive days. The device is a handheld electrical pulse generator and a pair of electrodes will be placed on the skin for stimulation. The electrical pulse generator is turned on and the amplitude of stimulation increased to the greatest amount tolerated. Patients will be followed through day 57 to assess durability of the intervention.
  Arms: Vagus Nerve Stimulation
Device: Sham vagus nerve stimulation — Patients will receive transcutaneous stimulation of the vagus nerve for 5 minutes daily for 28 consecutive days. The device is a handheld electrical pulse generator and a pair of electrodes will be placed on the skin for stimulation. The electrical pulse generator is turned on and the amplitude of stimulation increased to the greatest amount tolerated, however, the vagus nerve will not be stimulated. Patients will be followed through day 57 to assess durability of the intervention.
  Arms: Sham Vagus Nerve Stimulation

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic autoimmune inflammatory disease. Joint and muscle pain and fatigue are extremely common among patients and contribute to a reduced quality of life. Available therapies may be associated with significant side effects and many patients do not achieve an adequate response to these treatments. Therefore, there is an unmet need to develop new strategies to reduce pain and fatigue. Filling this need would significantly improve patients' quality of life. This trial will evaluate the effects of a novel approach, stimulating the vagus nerve, a nerve originating in the brain as a potential therapeutic intervention for treatment of musculoskeletal pain and fatigue. Vagus nerve stimulation has multiple beneficial effects and is one of the body's own ways to modulate the immune system. One can stimulate the vagus nerve via the skin at the neck or at specific locations in the ear, (transcutaneous vagus nerve stimulation: tcVNS). We recently completed a short, small scale randomized, placebo controlled trial of tcVNS in patients with SLE and observed dramatic benefits on musculoskeletal pain and fatigue. The treatment was safe without side effects. We are therefore proposing a longer trial to validate our initial findings and to look at durability. In this study, 18 patients with musculoskeletal pain will be followed for 2 months and will receive tcVNS or placebo (sham stimulation) for 5 minutes/day for 28 days. Patients will have a 1 out of 3 chance of receiving sham stimulation and neither the patient nor the evaluating investigator will know the actual treatment. The stimulations are self-administered, are non-painful and have not been associated with serious risks. After 28 days of stimulation, treatment will be discontinued and patients will be monitored for an additional 28 days to evaluate durability. Pain, fatigue and disease activity will be evaluated as well as possible side effects will be monitored throughout the trial. This study will also explore biologic mechanisms that may be responsible for the potential clinical effects. This will include possible effects of stimulation on gut permeability and the stool microbiome, areas that may play a significant role contributing to SLE disease and its manifestations. The development of an effective treatment without significant side effects would be extremely valuable and a significant advance for patients with SLE. If efficacious, tcVNS offers a non-toxic, non-immunosuppressive strategy to control two of the most common symptoms of this disease.

DETAILED DESCRIPTION:
Musculoskeletal (MS) pain and fatigue are common symptoms of patients with Systemic Lupus Erythematosus (SLE) affecting up to 95% and contributing to a reduced quality of life. Safe and efficacious treatment remains an unmet need for these disease manifestations. Stimulation of the vagus nerve results in beneficial effects in patients. We recently completed a short , small scale, randomized, sham-controlled, double blind clinical trial of transcutaneous vagus nerve stimulation (taVNS) in patients with SLE. The clinical benefit on MS pain and fatigue was dramatic. We now propose a randomized sham controlled clinical trial assessing the efficacy and durability of a longer exposure to taVNS (28 days in comparison to the 4 day exposure in the previous trial) in 18 patients randomized 2: 1 with musculoskeletal pain. After 28 days of stimulation, the treatment will be discontinued and patients will be monitored for an additional 28 days to evaluate the treatment's durability. Pain, fatigue, disease activity (global and musculoskeletal) and safety will be evaluated and safety will be monitored throughout the trial. In this clinical trial we will also explore potential biologic mechanisms and pathways by which taVNS exerts ifs effects in SLE, including potential effects on gut permeability and the microbiome.

ELIGIBILITY:
Inclusion Criteria:

* SLE (defined by the ACR or SLICC criteria),
* Musculoskeletal pain ≥ 4 on a non-anchored VAS 10 cm scale,
* BILAG C or greater on the Musculoskeletal Domain of the BILAG 2004,
* If on corticosteroids, the dose must be stable and ≤ 10 mg/day (prednisone or equivalent) for at least 14 days before baseline,
* If on background immunosuppressive treatment the dose must be stable for at least 28 days before baseline,
* If on NSAIDS, the dose must be stable for at least 7 days before baseline and the subject must be willing not to change the dose during the trial (except for toxicity),
* Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

* Initiation of immunosuppressive or antimalarial treatment within 3 months of baseline,
* Treatment with cyclophosphamide within 2 months of baseline,
* Initiation of anifrolumab within 3 months of baseline
* Initiation of belimumab within 6 months of baseline,
* Expectation to increase steroids and/or immunosuppressive treatment,
* Anti-phospholipid syndrome,
* Fibromyalgia,
* Treatment with an anti-cholinergic medication, including over the counter medications,
* Any implantable electronic devices including pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators,
* Current tobacco or nicotine user (to limit potential confounding effects of exposure to nicotine),
* Joint replacement within 60 days prior to study enrollment or planned within the course of the study,
* Any planned surgical procedure requiring general anesthesia within the course of the study,
* Intra-articular cortisone injections within 28 days of the start of study,
* Chronic inflammatory disorders apart from SLE affecting the joints,
* Investigational drug and/or treatment during the 28 days or seven half-lives of the investigational drug prior to the start of study drug dosing (Day 0), whichever is the greater length of time,
* Active infection including hepatitis B or hepatitis C at baseline,
* Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to a study intervention,
* Pregnancy or lactation (Pregnancy status will be determined via serum blood test & lactation will be determined via self-report),
* Comorbid disease that has previously required administration of corticosteroid use,
* Known allergy to mannitol or lactulose,
* Chronic treatment with narcotic medication,
* Prior receipt of transauricular vagus nerve stimulation in a clinical trial,
* Inability to comply with study and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Musculoskeletal Pain From Baseline. | 28 days
  Patients rate their musculoskeletal pain by making a mark on a 10cm anchored Visual Analog Scale where 0=no musculoskeletal pain and 10 =worst possible musculoskeletal pain.

SECONDARY OUTCOMES:
Percentage of Subjects With Treatment Emergent Adverse Events. | 57 days
  The percentage of participants with grade 2 or higher or specific grade 1 treatment emergent adverse events will be assessed using the NCI-CTAEversion4.
  The percentage of participants with grade 2 or higher treatment emergent adverse events will be assessed using the NCI-CTAEversion4.
  The percentage of participants with grade 2 or higher treatment emergent adverse events will be assessed using the NCI-CTAEversion4.
Change in Musculoskeletal Pain From Baseline | 5 days
  Patients rate their musculoskeletal pain by making a mark on a 10cm anchored Visual Analog Scale where 0=no musculoskeletal pain and 10 =worst possible musculoskeletal pain.
Change in Musculoskeletal Pain From Baseline | 57 days
  Patients rate their musculoskeletal pain by making a mark on a 10cm anchored Visual Analog Scale where 0=no musculoskeletal pain and 10 =worst possible musculoskeletal pain.
Change in Musculoskeletal Pain From Day 29 to Day 57 | day 29 to day 57
  Patients rate their musculoskeletal pain by making a mark on a 10cm anchored Visual Analog Scale where 0=no musculoskeletal pain and 10 =worst possible musculoskeletal pain.
Fatigue | 5 days
  Change from baseline fatigue will be measured using the FACIT F (Functional Assessment of Chronic Illness Therapy) questionnaire. The score ranges from 0 to 52, a higher score indicates less fatigue.
Fatigue | 28 days
  Change from baseline fatigue will be measured using the FACIT F (Functional Assessment of Chronic Illness Therapy) questionnaire. The score ranges from 0 to 52, a higher score indicates less fatigue.
Fatigue | 57 days
  Change from baseline fatigue will be measured using the FACIT F (Functional Assessment of Chronic Illness Therapy) questionnaire. The score ranges from 0 to 52, a higher score indicates less fatigue.
Fatigue | day 29 to day 57
  Change from Day 29 fatigue to Day 57 will be measured using the FACIT F (Functional Assessment of Chronic Illness Therapy) questionnaire. The score ranges from 0 to 52, a higher score indicates less fatigue.
Tender Joint Reduction | 5 days
  The percentage of tender joints reduced from baseline assessed by an investigator upon examining 68 potential tender joints.
Tender Joint Reduction | 28 days
  The percentage of tender joints reduced from baseline assessed by an investigator upon examining 68 potential tender joints.
Tender Joint Reduction | 57 days
  The percentage of tender joints reduced from baseline assessed by an investigator upon examining 68 potential tender joints.
Tender Joint Reduction | Day 29 to Day 57
  The percentage of tender joints reduced from day 29 to day 57 will be assessed by an investigator upon examining 68 potential tender joints.
Swollen joint reduction | 5 days
  The percentage of swollen joints reduced from baseline assessed by an investigator upon examining 66 potential swollen joints. Data shown for seven taVNS and five SS subjects with swollen joints at baseline.
Swollen joint reduction | 28 days
  The percentage of swollen joints reduced from baseline assessed by an investigator upon examining 66 potential swollen joints. Data shown for seven taVNS and five SS subjects with swollen joints at baseline.
Swollen joint reduction | 57 days
  The percentage of swollen joints reduced from baseline assessed by an investigator upon examining 66 potential swollen joints. Data shown for seven taVNS and five SS subjects with swollen joints at baseline.
Swollen joint reduction | Day 29 to Day 57
  The percentage of swollen joints reduced from Day 29 to Day 57 assessed by an investigator upon examining 66 potential swollen joints. Data shown for seven taVNS and five SS subjects with swollen joints at baseline.
Physician Global Assessment of Disease Activity (PGA) | Day 5
  Change in PGA from baseline, an anchored visual analog scale.ranging from 0 to 3 with higher scores signifying higher disease activity.
Physician Global Assessment of Disease Activity (PGA) | Day 28
  Change in PGA from baseline, an anchored visual analog scale.ranging from 0 to 3 with higher scores signifying higher disease activity.
Physician Global Assessment of Disease Activity (PGA) | Day 57
  Change in PGA from baseline, an anchored visual analog scale.ranging from 0 to 3 with higher scores signifying higher disease activity.
Physician Global Assessment of Disease Activity (PGA) | Days 29 to 57
  Change in PGA from day 29 to day 57; PGA is an anchored visual analog scale.ranging from 0 to 3 with higher scores signifying higher disease activity.
Patient Global Assessment of Disease (PtGA) | Day 5
  Change in PtGA from baseline, an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher disease activity.
Patient Global Assessment of Disease (PtGA) | Day 28
  Change in PtGA from baseline, an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher disease activity.
Patient Global Assessment of Disease (PtGA) | Day 57
  Change in PtGA from baseline, an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher disease activity.
Patient Global Assessment of Disease (PtGA) | Days 29 to 57
  Change in PtGA from day 29 to 57; PtGA is an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher disease activity.
Pain intensity | 5 days
  Pain intensity assessed by the PROMIS Pain Intensity Form 1a which asks subjects to mark a scale rating the average pain intensity over the past 7 days. The rating scale consists of whole numbers from 1 to 10. The PROMIS Pain Intensity Scale is a series of 3 questions that assess pain intensity at its worst, at its average, and at current moment. A higher score indicates higher levels of pain intensity.
Pain intensity | 28 days
  Pain intensity assessed by the PROMIS Pain Intensity Form 1a which asks subjects to mark a scale rating the average pain intensity over the past 7 days. The rating scale consists of whole numbers from 1 to 10. The PROMIS Pain Intensity Scale is a series of 3 questions that assess pain intensity at its worst, at its average, and at current moment. A higher score indicates higher levels of pain intensity.
Pain intensity | 57 days
  Pain intensity assessed by the PROMIS Pain Intensity Form 1a which asks subjects to mark a scale rating the average pain intensity over the past 7 days. The rating scale consists of whole numbers from 1 to 10. The PROMIS Pain Intensity Scale is a series of 3 questions that assess pain intensity at its worst, at its average, and at current moment. A higher score indicates higher levels of pain intensity.
Pain intensity | Days 29 to 57
  Pain intensity assessed by the PROMIS Pain Intensity Form 1a which asks subjects to mark a scale rating the average pain intensity over the past 7 days. The rating scale consists of whole numbers from 1 to 10. The PROMIS Pain Intensity Scale is a series of 3 questions that assess pain intensity at its worst, at its average, and at current moment. A higher score indicates higher levels of pain intensity.
Pain interference | 5 days
  Pain interference will be assessed by requesting subjects to answer the PROMIS Pain Interference Short Form 8a. The PROMIS Pain Interference Short Form 8a is a series of 8 questions which asks how much has pain interfered with different aspects of activities of daily living over the previous 7 days
Pain interference | 28 days
  Pain interference will be assessed by requesting subjects to answer the PROMIS Pain Interference Short Form 8a. The PROMIS Pain Interference Short Form 8a is a series of 8 questions which asks how much has pain interfered with different aspects of activities of daily living over the previous 7 days
Pain interference | 57 days
  Pain interference will be assessed by requesting subjects to answer the PROMIS Pain Interference Short Form 8a. The PROMIS Pain Interference Short Form 8a is a series of 8 questions which asks how much has pain interfered with different aspects of activities of daily living over the previous 7 days
Pain interference | Days 29 to 57
  Pain interference will be assessed by requesting subjects to answer the PROMIS Pain Interference Short Form 8a. The PROMIS Pain Interference Short Form 8a is a series of 8 questions which asks how much has pain interfered with different aspects of activities of daily living over the previous 7 days
Health Related Quality of Life (HRQoL)) | 28 days
  HRQoL will be evaluated using the LupusQoL, a validated SLE specific index which assesses 8 domains including physical health, emotional health, body image, pain, planning, fatigue, intimate relationships, and burden to others. Higher scores correspond to worse quality-of-life.
Health Related Quality of Life (HRQoL)) | Day 57
  HRQoL will be evaluated using the LupusQoL, a validated SLE specific index which assesses 8 domains including physical health, emotional health, body image, pain, planning, fatigue, intimate relationships, and burden to others. Higher scores correspond to worse quality-of-life.
Health Related Quality of Life (HRQoL)) | Days 29 to 57
  HRQoL will be evaluated using the LupusQoL, a validated SLE specific index which assesses 8 domains including physical health, emotional health, body image, pain, planning, fatigue, intimate relationships, and burden to others. Higher scores correspond to worse quality-of-life.
Anxiety | Day 29
  Promis Anxiety Short Form will assess anxiety. It is an 8 item questionaire assessing components related to anxiety including fear, anxious misery, hyperarousal, and somatic symptoms. Higher scores indicate greater levels of anxiety.
Anxiety | Day 57
  Promis Anxiety Short Form will assess anxiety. It is an 8 item questionaire assessing components related to anxiety including fear, anxious misery, hyperarousal, and somatic symptoms. Higher scores indicate greater levels of anxiety.
Anxiety | Days 29 to 57
  Promis Anxiety Short Form will assess anxiety. It is an 8 item questionaire assessing components related to anxiety including fear, anxious misery, hyperarousal, and somatic symptoms. Higher scores indicate greater levels of anxiety.
Depression | Day 28
  Beck Depression Inventory (BDI) will assess depression. The BDI is a 21 item questionnaire measuring the severity of depression. Higher scores indicate greater levels of depression.
Depression | Day 57
  Beck Depression Inventory (BDI) will assess depression. The BDI is a 21 item questionnaire measuring the severity of depression. Higher scores indicate greater levels of depression.
Depression | Days 29 to 57
  Beck Depression Inventory (BDI) will assess depression. The BDI is a 21 item questionnaire measuring the severity of depression. Higher scores indicate greater levels of depression.
Polysymptomatic distress | Day 29
  Polysymptomatic distress will be assessed by the Fibromyalgia Symptom Score (FSS), a patient reported outcome measuring the extent of polysymptomatic distress on a scale ranging from 0-31. Higher scores correspond to greater polysymptomatic distress.
Polysymptomatic distress | Day 57
  Polysymptomatic distress will be assessed by the Fibromyalgia Symptom Score (FSS), a patient reported outcome measuring the extent of polysymptomatic distress on a scale ranging from 0-31. Higher scores correspond to greater polysymptomatic distress.
Polysymptomatic distress | Days 29 to 57
  Polysymptomatic distress will be assessed by the Fibromyalgia Symptom Score (FSS), a patient reported outcome measuring the extent of polysymptomatic distress on a scale ranging from 0-31. Higher scores correspond to greater polysymptomatic distress.
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2K) | Day 28
  SLEDAI-2K is a 24 item index which are scored by an investigator as either present or absent. Items include clinical and laboratory features of SLE. Higher scores correspond to greater disease activity.
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2K) | Day 57
  SLEDAI-2K is a 24 item index which are scored by an investigator as either present or absent. Items include clinical and laboratory features of SLE. Higher scores correspond to greater disease activity.
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI-2K) | Days 29 to 57
  SLEDAI-2K is a 24 item index which are scored by an investigator as either present or absent. Items include clinical and laboratory features of SLE. Higher scores correspond to greater disease activity.
BILAG (British Isles Lupus Assessment Group) 2004 | Day 28
  BILAG 2004 index assesses SLE disease activity in nine organ symptoms. Each domain is categorized into 1 of 5 levels (A, B, C, D, E). Lower letters (e.g. A) indicate more active disease.
BILAG (British Isles Lupus Assessment Group) 2004 | Day 57
  BILAG 2004 index assesses SLE disease activity in nine organ symptoms. Each domain is categorized into 1 of 5 levels (A, B, C, D, E). Lower letters (e.g. A) indicate more active disease.
BILAG (British Isles Lupus Assessment Group) 2004 | Days 29 to 57
  BILAG 2004 index assesses SLE disease activity in nine organ symptoms. Each domain is categorized into 1 of 5 levels (A, B, C, D, E). Lower letters (e.g. A) indicate more active disease.
CLASI (Cutaneous LE Disease Area and Severity Index) | Day 28
  CLASI assesses SLE skin disease activity and damage. Higher scores indicate greater levels of cutaneous disease.
CLASI (Cutaneous LE Disease Area and Severity Index) | Day 57
  CLASI assesses SLE skin disease activity and damage. Higher scores indicate greater levels of cutaneous disease.
CLASI (Cutaneous LE Disease Area and Severity Index) | Days 29 to 57
  CLASI assesses SLE skin disease activity and damage. Higher scores indicate greater levels of cutaneous disease.
Musculoskeletal disease activity--patient | Day 5
  Musculoskeletal disease activity will be assessed by patients by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher musculoskeletal disease activity.
Musculoskeletal disease activity--patient | Day 29
  Musculoskeletal disease activity will be assessed by patients by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher musculoskeletal disease activity.
Musculoskeletal disease activity--patient | Day 57
  Musculoskeletal disease activity will be assessed by patients by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher musculoskeletal disease activity.
Musculoskeletal disease activity--patient | Days 29 to 57
  Musculoskeletal disease activity will be assessed by patients by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher musculoskeletal disease activity.
Musculoskeletal disease activity--physician | Day 5
  Musculoskeletal disease activity will be assessed by the physician investigator by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher musculoskeletal disease activity.
Musculoskeletal disease activity--physician | Day 28
  Musculoskeletal disease activity will be assessed by the physician investigator by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher musculoskeletal disease activity.
Musculoskeletal disease activity--physician | Day 57
  Musculoskeletal disease activity will be assessed by the physician investigator by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher musculoskeletal disease activity.
Musculoskeletal disease activity--physician | Days 28 to 57
  Musculoskeletal disease activity will be assessed by the physician investigator by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying higher musculoskeletal disease activity.
Morning Stiffness | Day 5
  Morning stiffness will be assessed by patients by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying greater morning stiffness.
Morning Stiffness | Day 28
  Morning stiffness will be assessed by patients by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying greater morning stiffness.
Morning Stiffness | Day 57
  Morning stiffness will be assessed by patients by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying greater morning stiffness.
Morning Stiffness | Days 29 to 57
  Morning stiffness will be assessed by patients by an anchored visual analog scale.ranging from 0 to 10 with higher scores signifying greater morning stiffness.
Patient assessment of response | Day 5
  Patient assessment of response will be determined by a 5 component Likert scale by the patient.
Patient assessment of response | Day 28
  Patient assessment of response will be determined by a 5 component Likert scale by the patient.
Patient assessment of response | Day 57
  Patient assessment of response will be determined by a 5 component Likert scale by the patient.
Physician assessment of response | Day 5
  Patient assessment of response will be determined by a 5 component Likert scale by the physician investigator.
Physician assessment of response | Day 28
  Patient assessment of response will be determined by a 5 component Likert scale by the physician investigator.
Physician assessment of response | Day 57
  Patient assessment of response will be determined by a 5 component Likert scale by the physician investigator.
Lupus Low Disease Activity State (LLDAS) | Day 28
  LLDAS is a state achieved when there are minimal signs or symptoms of lupus disease activity while the patient is on low dose corticosteroids and stable therapy.
Lupus Low Disease Activity State (LLDAS) | Day 57
  LLDAS is a state achieved when there are minimal signs or symptoms of lupus disease activity while the patient is on low dose corticosteroids and stable therapy.
SRI-4 | Day 28
  SRI-4 is a composite categorical response measure of improvement in SLE disease activity from a comparator timepoint/baseline. Achievement of the SRI-4 indicates a clinically meaningful response.
SRI-4 | Day 57
  SRI-4 is a composite categorical response measure of improvement in SLE disease activity from a comparator timepoint/baseline. Achievement of the SRI-4 indicates a clinically meaningful response.

OTHER OUTCOMES:
Functional gut permeability | Day 28
  Functional gut permeability is assessed by measuring urinary C mannitol/lactulose ratios after oral injestion of the sugars, in timed urine collections over 24 hours.
Stool microbiome | Day 28
  Stool microbiome is assessed by determining changes in metagenomics, metatranscriptomics and metabolomics from baseline in stool specimens.
Gut permeability: serum I-FABP, zonulin and LPS, and by stool calprotectin and zonulin | Day 28
  Gut permeability: serum I-FABP is determined by measuring levels of serum I-FABP
Gut permeability: zonulin | Day 28
  Gut permeability: zonulin is determined by measuring levels of serum zonulin
Gut permeability: Lipopolysaccharide (LPS) | Day 28
  Gut permeability: Lipopolysaccharide (LPS) is determined by measuring levels of serum LPS.
Gut permeability: Stool calprotectin | Day 28
  Gut permeability: Stool calprotectin is determined by measuring levels of calprotectin in the stool.
Gut permeability: Stool zonulin | Day 28
  Gut permeability: Stool zonulin is determined by measuring levels of zonulin in the stool.
Oxidative stress | Day 28
  Oxidative stress is determined by measuring levels of circulating glutathione and oxidized glutathione
Oxidative stress | Day 57
  Oxidative stress is determined by measuring levels of circulating glutathione and oxidized glutathione
Neurotrophins | Day 28
  Neurotrophins are determined by measuring circulating levels of neurotrophins (nerve growth factor (NGF) and brain-derived neurotrophic factor (BDNF).
Neurotrophins | Day 57
  Neurotrophins are determined by measuring circulating levels of neurotrophins (nerve growth factor (NGF) and brain-derived neurotrophic factor (BDNF).
Neurotrophins | Days 29 to 57
  Neurotrophins are determined by measuring circulating levels of neurotrophins (nerve growth factor (NGF) and brain-derived neurotrophic factor (BDNF).
Kynurenine pathway metabolites | Day 28
  Kynurenine pathway metabolites are determined by measuring circulating levels of tryptophan, kynurenine, kynurenic acid and quinolinic acid
Kynurenine pathway metabolites | Day 57
  Kynurenine pathway metabolites are determined by measuring circulating levels of tryptophan, kynurenine, kynurenic acid and quinolinic acid
Kynurenine pathway metabolites | Days 28 to 57
  Kynurenine pathway metabolites are determined by measuring circulating levels of tryptophan, kynurenine, kynurenic acid and quinolinic acid
Neuropeptides | Day 28
  Neuropeptides are determined by measuring circulating levels of substance P, calcitonin gene-related peptide (CGRP) and neuropeptide Y (NPY), neuropeptide B (NPB) and neuropeptide W (NPW).
Neuropeptides | Day 57
  Neuropeptides are determined by measuring circulating levels of substance P, calcitonin gene-related peptide (CGRP) and neuropeptide Y (NPY), neuropeptide B (NPB) and neuropeptide W (NPW).
Neuropeptides | Days 29 to 57
  Neuropeptides are determined by measuring circulating levels of substance P, calcitonin gene-related peptide (CGRP) and neuropeptide Y (NPY), neuropeptide B (NPB) and neuropeptide W (NPW).
Erythrocyte Sedimentation Rate (ESR) | Day 5
  ESR is a laboratory parameter reflecting inflammation. It measures the rate that erythrocytes sediment (fall) over a specific period of time.
Erythrocyte Sedimentation Rate (ESR) | Day 28
  ESR is a laboratory parameter reflecting inflammation. It measures the rate that erythrocytes sediment (fall) over a specific period of time.
Erythrocyte Sedimentation Rate (ESR) | Day 57
  ESR is a laboratory parameter reflecting inflammation. It measures the rate that erythrocytes sediment (fall) over a specific period of time.
Erythrocyte Sedimentation Rate (ESR) | Days 28 to 57
  ESR is a laboratory parameter reflecting inflammation. It measures the rate that erythrocytes sediment (fall) over a specific period of time.
Complement component 3 (C3) | Day 28
  Serum levels of C3 are measured in a clinical laboratory
Complement component 3 (C3) | Day 57
  Serum levels of C3 are measured in a clinical laboratory
Complement component 3 (C3) | Days 28 to 57
  Serum levels of C3 are measured in a clinical laboratory
Complement component 4 (C4) | Day 28
  Serum levels of C4 are measured in a clinical laboratory
Complement component 4 (C4) | Day 57
  Serum levels of C4 are measured in a clinical laboratory
Complement component 4 (C4) | Days 28 to 57
  Serum levels of C4 are measured in a clinical laboratory
Anti-DNA antibodies | Day 28
  Serum levels of anti-DNA antibodies are measured by a laboratory
Anti-DNA antibodies | Day 57
  Serum levels of anti-DNA antibodies are measured by a laboratory
Anti-DNA antibodies | Days 28 to 57
  Serum levels of anti-DNA antibodies are measured by a laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aranow, MD, Principal Investigator — Northwell Health

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with researchers with a proposals directed to caranow@northwell.edu. IPD data collected during the trial, after deidentification hat underlie results in a publication will be shared and will be available by 6 months to 3 years following publication of the manuscript.
  gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website
Supporting Information: CSR
Time Frame: 6 months to 3 years after publication
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal and/or whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.